CLINICAL TRIAL: NCT01018199
Title: Use of Procalcitonin (PCT) and C-reactive Protein (CRP) to Guide Antibiotic Therapy in Community Acquired Pneumonia: a Randomized Controlled Trial
Brief Title: Procalcitonin Versus C-reactive Protein to Guide Therapy in Community Acquired Pneumonia
Acronym: CAP-Marker
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in the profile of patients assisted by the hospital
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Vandack Alencar Nobre, Associate Professor, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFMG-PCT
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2012-03

CONDITIONS: Community-acquired Pneumonia
Keywords: C-reactive protein; procalcitonin; community-acquired pneumonia; antibiotic therapy
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1- C-reactive protein (CRP) guided antibiotic therapy (Experimental): Intervention on antibiotic therapy will be based on circulating RCP levels
  Interventions: Other: CRP
- Group 2 - procalcitonin (PCT) guided antibiotic therapy (Active Comparator): Intervention on antibiotic therapy will be based on circulating PCT levels
  Interventions: Other: PCT

INTERVENTIONS:
Other: CRP — C-reactive protein guided antibiotic therapy plasma CRP measurement to guide the duration of antibiotic therapy
  Arms: Group 1- C-reactive protein (CRP) guided antibiotic therapy
Other: PCT — Procalcitonin guided antibiotic therapy plasma PCT measurement to guide the duration of antibiotic therapy
  Arms: Group 2 - procalcitonin (PCT) guided antibiotic therapy

SUMMARY:
In this study the investigators aim to test if C-reactive protein (CRP) or procalcitonin(PCT) - guided strategy allows to reduce the antibiotic use in patients wiht community-acquired pneumonia. Therefore, the safety of this intervention will be carefully measured.

DETAILED DESCRIPTION:
Methods

• Patients and settings:

All adult (> 18 years old) patients with diagnosis community-acquired pneumonia will receive initial antibiotic therapy based on local guidelines and susceptibility patterns, according to the decision of the treating physician.Patients will be randomly assigned to one of two groups, which respectively include PCR and PCT clinical procedure protocol. Randomization will be done using a table of random numbers generated by computer. For practical reasons the doctors treating the patients in question have science group in which the patient was included.

Patients included in the two groups will have baseline assessment during the first day of study:

* Clinical evaluation of basic
* Start of antibiotic therapy
* Inclusion in the study
* Randomization (after signing the Informed Consent)
* Interventions:

They will have circulating PCT and CRP levels measured at baseline and days 1,2,3 e 5 in both groups.

Group 1 - CRP group: the duration of antibiotic therapy will be based on circulating CRP levels.

Group 2 - PCT group: the duration of antibiotic therapy will be based on circulating PCT levels.

Patients enrolled in the study will undergo daily measurements of plasma CRP (Dry Chemistry - Johnsons & Johnsons) and PCT (BRAHMS PCT VIDAS) levels up to day 5, and then, every 48hr in patients remaining in the ICU, and every 5 days in those transferred to the ward. Patients will be followed up 28 days, or until death or hospital transference, which comes first. PCT and CRP results will be released in sealed envelopes. During the study period, only the results corresponding to the patient randomization group will be open; i.e., CRP for CRP group patients and PCT for PCT group patients.

Criteria for antibiotic interruption:

The investigators will propose the interruption of antibiotics if:

1. The patients is clinically stable, without signs of active infection
2. CRP group: a relative reduction of 50% in baseline CRP levels, or a value lower than 25mg/dl is reached.
3. PCT group: a relative reduction of 90% in baseline PCT levels, or if a absolute value lower than 0.1 ng/ml is reached.

The final decision regarding antibiotic therapy will be always let to the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Signed informed consent
3. Suspected or confirmed community-acquired pneumonia

Exclusion Criteria:

1. Nosocomial pneumonia: development of symptoms after 48 hours of admission to the Emergency Department, or within 14 days after hospital discharge
2. Patients with lung cancer confirmed strongly suspected.
3. Patients with severe immunosuppression, such as severe neutropenia (<500 neutrófilos/mm3), use of corticosteroids in doses above 0.5 mg / kg / day of prednisone or equivalent for at least 2 weeks, transplantation of solid organs or cells hematopoietic, use of immunosuppressants for any other reason (eg. azathioprine or cyclosporine), hipogamagloulinemia
4. Patients with asplenia in any order
5. Pregnant
6. Patients with known HIV infection
7. Stay indicated only for social reasons
8. Patients on antibiotics for any other reason
9. Patients with multiple trauma, burns or surgery grid size in the last 5 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Duration of antibiotic therapy for the first episode of infection | 28 days
Total antibiotic exposure days per 1,000 days | 28 days
Days alive without antibiotics | 28 days

SECONDARY OUTCOMES:
All cause 28-day mortality | 28 days
clinical cure rate | 28 days
Infection relapse (diagnosed less than 48h after antibiotic discontinuation) | 28 days
Length of hospitalization stay | Whole hospitalization
In-hospital mortality | 28 days
Nosocomial infection rate | 28 days
Nosocomial superinfection (diagnosed more than 48hous after discontinuation of the antibiotic therapy given to the first episode of infection) | 28 days
Isolation of resistant bacteria | 28 days
All cause 90-day mortality | 90 days
costs of hospitalization | Whole hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Vandack A Nobre, PhD, Principal Investigator — Medical School of the Federal University of Minas Gerais; Karla F Finotti, MD, Study Chair — Medical School of the Federal University of Minas Gerais
Locations (1):
- Hospital das Clínicas - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided